CLINICAL TRIAL: NCT06504901
Title: Evaluation of Efficacy and Safety of PD-1 Monoclonal Antibody in Combination With rhG-CSF, IL-2, and CapeOX in Initially Resectable Synchronous Colorectal Liver Metastases: A Single-Center, Single-Arm, Open-Label Clinical Study (PRICE)
Brief Title: Evaluation of Efficacy and Safety of PD-1 Monoclonal Antibody in Combination With rhG-CSF, IL-2, and CapeOX in Initially Resectable Synchronous Colorectal Liver Metastases
Status: Not yet recruiting | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: PRICE202407
Record Dates: First submitted 2024-07-11; First posted 2024-07-17 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Colorectal Cancer
Keywords: Tislelizumab; Interleukin-2; MSS/pMMR colorectal cancer; rhG-CSF
MeSH Terms: conditions — Colorectal Neoplasms | interventions — tislelizumab; Interleukin-2; Capecitabine; Oxaliplatin; Filgrastim

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CapeOX+PD-1+IL-2+rhG-CSF: Tislelizumab 200mg ivd D1 + Interleukin 2 100IU HD,QOD d1-d14+rhG-CSF 5mcg/kg HD, QD d1-d14 +CapeOX (Capecitabine: 1000mg/m2 bid po, d1-d14；Oxaliplatin 130mg/m2 ivd, d1) 6 cycles
  Interventions: Drug: Tislelizumab; Drug: Interleukin-2; Drug: Capecitabine; Drug: Oxaliplatin; Drug: Neupogen

INTERVENTIONS:
Drug: Tislelizumab — Tislelizumab 200mg ivd D1
Drug: Interleukin-2 — Interleukin 2 100IU HD,QOD d1-d14
Drug: Capecitabine — Capecitabine: 1000mg/m2 bid po, d1-d14
Drug: Oxaliplatin — Oxaliplatin 130mg/m2 ivd, d1
Drug: Neupogen — rhG-CSF 5mcg/kg HD, QD d1-d14

SUMMARY:
This study attempts to employ a combination therapy using rhG-CSF, IL-2, and PD-1 inhibitors, aiming to overcome the limitations of monotherapy in immunotherapy through multi-faceted immune regulation. By modulating the immune microenvironment to enhance immune cell infiltration, and breaking through the physical and immunosuppressive barriers of tumors, it seeks to augment the efficacy of immunotherapy. This approach explores the effectiveness of a neoadjuvant treatment model in cases of liver metastasis.

DETAILED DESCRIPTION:
Colorectal cancer stands as a prominent global health issue, ranking among the most prevalent malignancies worldwide. Its incidence exhibits distinct geographical variations, with higher rates observed in developed countries. Age is a significant risk factor, primarily affecting individuals aged 50 and above, although a concerning trend of increasing incidence in younger adults has emerged in recent years. There exists a gender disparity, with a slightly higher prevalence in males. Notably, lifestyle factors, including dietary choices, sedentary habits, smoking, and obesity, play pivotal roles in its pathogenesis. These epidemiological patterns underscore the urgency of implementing effective prevention strategies and advancing early detection methods to mitigate the impact of the disease.

The poor prognosis in colorectal cancer patients primarily stems from the tumor's aggressive biological properties and its propensity for distant metastasis. The unique anatomy of the liver, endowed with both the portal venous and hepatic arterial systems, and abundant blood supply, renders it the most common site for distant metastasis from colorectal cancer. Currently, radical surgical resection remains the primary treatment for colorectal liver metastases; however, due to tumor burden and clinical complications, only 17% to 20% of patients with colorectal liver metastases are amenable to surgery. With advancements in therapeutic modalities and the precision of medical approaches, a comprehensive treatment paradigm combining surgery, radiofrequency ablation, postoperative targeted drugs, and interventional therapies has gradually taken shape. Although this has enriched treatment options for colorectal liver metastases and improved outcomes, many patients present with multifocal intrahepatic metastases and severe complications at diagnosis, precluding further surgical intervention and resulting in limited survival and poor prognosis. In recent years, immunotherapy for tumors has garnered unprecedented attention and extensive clinical application, fundamentally relying on enhancing the patient's own immune capabilities to bolster antitumor activity. The ongoing in-depth investigation into the programmed cell death receptor 1 (PD1)/programmed cell death ligand 1 (PDL1) signaling pathway has also presented new opportunities for patients with colorectal liver metastases.

In colorectal cancer, the PD-1 inhibitory pathway plays a central role in regulating immune cell exhaustion. However, a majority of colorectal cancer patients exhibit limited response to monotherapy targeting PD-1, suggesting that combinations of PD1 inhibitors with other immunostimulatory agents may address this challenge. Some of these combination therapies have made progress in animal models and are being tested in clinical studies. Among them, interleukin-2 (IL-2) emerges as a promising candidate to synergize with PD-1 blockade in exerting antitumor effects. Meanwhile, recombinant human granulocyte colony-stimulating factor (rhG-CSF) has been primarily utilized in oncology for two purposes: first, to prevent and treat neutropenia induced by chemotherapy or radiotherapy; second, as a priming strategy to augment the efficacy of chemotherapy. Our study aims to explore a combination therapy employing rhG-CSF, IL-2, and PD-1 inhibitors, with the objective of overcoming the limitations of single-agent immunotherapy through multifaceted immune modulation. By modulating the immune microenvironment to enhance immune cell infiltration and breach the physical and immunosuppressive barriers of tumors, we seek to potentiate the effects of immunotherapy and investigate the efficacy of a neoadjuvant treatment model in liver metastases.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years and ≤75 years
2. Histologically confirmed colorectal adenocarcinoma
3. pMMR (proficient mismatch repair) or MSI-L (microsatellite instability-low) or MSS (microsatellite stable)
4. Synchronous liver metastases
5. Achievable NED (No Evidence of Disease) status
6. CRS (Clinical Risk Score) of 3-4 points
7. ECOG (Eastern Cooperative Oncology Group) Performance Status score ≤ 1

Exclusion Criteria:

1. Recurrent colorectal cancer with active bleeding, perforation, or complex conditions requiring urgent surgery; or concurrent non-colorectal cancer malignancies.
2. Patients who have previously received systemic anticancer therapy for colorectal cancer; or have been treated with PD-1, PD-L1, or CTLA-4 antibodies.
3. Patients with any active autoimmune disease; known or tested positive for Human Immunodeficiency Virus (HIV) or Acquired Immunodeficiency Syndrome (AIDS); or a history requiring steroid or immunosuppressive drug treatment.
4. Patients with interstitial lung disease, non-infectious pneumonitis, or uncontrolled systemic diseases (such as diabetes, hypertension, pulmonary fibrosis, and acute pneumonia).
5. Patients who experienced any Grade 2 or higher toxicities due to prior treatments (as classified by the Common Terminology Criteria for Adverse Events [CTCAE] version 5), which have not resolved (excluding anemia, alopecia, and skin pigmentation changes); known or suspected history of hypersensitivity to any of the drugs used in the trial.
6. Pregnant or breastfeeding women.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. Age ≥18 years and ≤75 years
  2. Histologically confirmed colorectal adenocarcinoma
  3. pMMR (proficient mismatch repair) or MSI-L (microsatellite instability-low) or MSS (microsatellite stable)
  4. Synchronous liver metastases
  5. Achievable NED (No Evidence of Disease) status
  6. CRS (Clinical Risk Score) of 3-4 points
  7. ECOG (Eastern Cooperative Oncology Group) Performance Status score ≤ 1
Sampling Method: Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2024-07-10 (Estimated); Primary Completion 2025-07-10 (Estimated); Study Completion 2027-07-10 (Estimated)

PRIMARY OUTCOMES:
CR rate (cCR + local excision pCR) | 3 years
  Complete Response rate," which includes both "complete clinical response" (cCR)

SECONDARY OUTCOMES:
Event-Free Survival rates | 5 years
  Event-Free Survival (EFS) is the length of time after treatment during which the patient survives without any events of interest occurring, such as disease progression, recurrence, or death. Therefore, the 1/2/3-year EFS rates refer to the percentages of patients surviving without these events at 1, 2, and 3 years.
Overall Survival rates | 5 years
  Overall Survival (OS) is the most common endpoint in cancer clinical trials, measuring the proportion of patients still alive at specific time points after the start of treatment. Thus, the 1/2/3-year OS rates represent the percentages of patients still alive at 1, 2, and 3 years post-treatment.

IPD SHARING:
Plan to Share IPD: Undecided